CLINICAL TRIAL: NCT04443036
Title: Albumin-bound Paclitaxel Combined With Toripalimab as First-line/Second-line Treatment of Local Advanced or Metastatic Gastric or Gastroesophageal Junction Carcinoma: A Prospective, Open-label, Single-arm Phase II Clinical Study
Brief Title: Clinical Study of Nab-paclitaxel Combined With Toripalimab in Local Advanced or Metastatic G/GEJ Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director of Department of Medical Oncology, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-ATJogress
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Gastric Carcinoma
Keywords: gastric carcinoma; gastroesophageal junction carcinoma; Albumin Bound Paclitaxel; Toripalimab
MeSH Terms: conditions — Stomach Neoplasms | interventions — Albumin-Bound Paclitaxel; Taxes; Paclitaxel; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Albumin-bound Paclitaxel Combined With Toripalimab (Experimental): * Albumin-bound Paclitaxel：125mg/m2 IV d1、8，Q3W
  * Toripalimab：240 mg，IV d1，Q3W
  * until disease progression, lost follow-up visit, death , unacceptable toxicity, Maximum treatment duration of Toripalimab is 24 months
  Interventions: Drug: Albumin-Bound Paclitaxel; Drug: Toripalimab

INTERVENTIONS:
Drug: Albumin-Bound Paclitaxel — * 125mg/m2 IV d1、8，Q3W
  * until disease progression, lost follow-up visit, death , unacceptable toxicity
  Other Names: Paclitaxel (albumin-bound); Paclitaxel for injection(Albumin Bound)
Drug: Toripalimab — * 240 mg，IV d1，Q3W
  * until disease progression, lost follow-up visit, death , unacceptable toxicity, Maximum treatment duration is 24 months

SUMMARY:
This study is to evaluate the efficacy and safety of Albumin-bound paclitaxel combined with Toripalimab as first-line/second-line treatment of local advanced or metastatic gastric or gastroesophageal junction carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-70 years old, female or male.
* Histopathologically diagnosed local advanced or metastatic gastric or gastroesophageal junction carcinoma, HER2 negative.
* At least one measurable lesion according to RECIST 1.1.
* ≤1 prior line. adjuvant/neoadjuvant therapy is allowed, adjuvant/neoadjuvant therapy is considered as the first-line treatment for advanced diseases, if recurrence occurs during the treatment or within 6 months after the last treatment. prior chemotherapy combined with targeted therapy is allowed.
* ECOG performance status of 0 or 1.
* Adequate organ and bone marrow function: ANC≥1.5×109/L, PLT≥90×109/L, HGB≥90g/L,TBil≤1.5ULN, ALT≤2.5ULN, AST≤2.5ULN, Serum Cr≤1ULN, endogenous creatinine clearance>60ml/min (Cockcroft-Gault formula).
* The international normalized ratio (INR) ≤ 1.5 and some prothrombin time (PPT or APTT) ≤ 1.5ULN within 7 days before enrollment.
* Expected survival≥3 months.
* Signed informed consent (ICF) before enrollment.
* Women of childbearing age must undergo a pregnancy test within 7 days prior to enrollment and have a negative result and are willing to use effective and reliable contraceptive methods during and 6 months after the last treatment.

Exclusion Criteria:

* History of severe allergic reactions to chimeric or humanized antibodies or fusion proteins, or known allergic to any component of Toripalimab or any component of Albumin Bound paclitaxel.
* severe hypersensitivity after previous administration of monoclonal antibody.
* ≥1 prior line therapy after progression.
* Prior therapy with PD-1、PD-L1/L2、CTLA-4 antibody, or any other immunotherapy.
* A history of organ transplantation.
* Any other malignancy within 5 years excluding healed Basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of cervical or breast.
* Received anti-tumor vaccine or other immune-stimulating agents (interferon, interleukin, thymosin, immuno cell therapy, etc.) within 1 month before the first treatment.
* Symptomatic central nervous system metastases.
* Acute or chronic Active hepatitis B or hepatitis C.
* Interstitial pneumonia, pneumoconiosis, drug-induced pneumonia, pulmonary fibrosis, severely impaired lung function and other pulmonary diseases.
* Active tuberculosis, receiving anti-TB treatment or have received anti-TB treatment within 1 year prior to first treatment.
* Human immunodeficiency virus (HIV) infection（HIV antibody positive）, or known syphilis infection.
* Severe uncontrolled disease, non-metastatic systemic disease, active or poor clinical control infection.
* Patients with autoimmune diseases or abnormal immune system.
* Treatment with immunosuppressive medications within 4 weeks prior to enrollment. Nasal spray, inhalation, or other ways of topical corticosteroids or systemic corticosteroids at physiologic doses （not to exceed 10 mg/day of prednisone or its equivalent Steroids）are not included.
* Expected to require any other form of antitumor therapy while on study (including maintenance therapy with any other drugs for gastric or gastroesophageal junction carcinoma、radiotherapy and/or surgical resection)
* Received major surgery or radiation therapy of > 30 Gy not to chest within 4 weeks of the first treatment, or radiation therapy of > 30 Gy to chest within 24 weeks of the first treatment,or radiation therapy of < 30 Gy to chest within 2 weeks of the first treatment, and had not recovered from the toxicity and/or complications of the most recent prior chemotherapy to Grade 1 or less (except alopecia or fatigue).
* Poorly Controlled Diabetes（fasting blood-glucose ≥CTCAE grade 2）.
* Clinically significant thyroid dysfunction and can't maintain thyroid hormone levels in the normal range with drugs.
* Use of any live vaccines within 4 weeks before enrollment.
* Pregnant or lactating subjects.
* Participated in any other drug clinical study within 4 weeks before the enrollment.
* Any other disease、metabolic disorders、Physical examination or laboratory abnormalities that might result in contraindications in the use of experimental drugs or affect the reliability of the study, or Puts patients at high risk.
* The investigator believes are not suitable for participating in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 24 months
  * Progression-Free Survival
  * Defined as the time from first dose of study medication to the first documented disease progression per RECIST version 1.1，or death from any cause, whichever occurred first

SECONDARY OUTCOMES:
ORR | up to 24 months
  * Objective Response Rate
  * Defined as the proportion of patients with confirmed complete response /partial response per RECIST version 1.1
DCR | up to 24 months
  * Disease control rate
  * Defined as the proportion of patients with confirmed complete response /partial response/ Stable Disease per RECIST version 1.1
OS | up to 24 months
  * Over survival
  * Defined as the time from the date of first dose of study medication to the date of death from any cause
Change in Quality of Life(QoL)：measured by EORTC QLQ-C30 questionnaire | up to 24 months
  * European Organisation for Research and Treatment of Cancer's Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
  * The change in the quality of life as measured by EORTC QLQ-C30, consists of 30 questions that provide a global QoL scale, five functional scales (physical, role-playing, emotional, cognitive, social), three symptom scales (fatigue, nausea and vomiting, pain) and six individual factors (dyspnea, insomnia, loss of appetite, constipation, diarrhea, financial difficulties). The scores of each scale are calculated in a score ranging from 0 to 100. A high score on a functional scale represents a good level of function.
Adverse events | up to 24 months
  - Defined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, PhD., Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China